CLINICAL TRIAL: NCT01480700
Title: Effect of Consumption of Eggs Rich in Xanthophyll Carotenoids and Omega-3 Fatty Acids on the Macular Pigment in Healthy People
Brief Title: Consumption of Eggs Rich in Lutein and Omega-3 Fatty Acids on the Macular Pigment
Acronym: ALGOVUE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur de Lille (Other)
Collaborators: Roquette Freres (Industry); Sanders (Unknown)
Responsible Party: Principal Investigator, Jean-Michel Lecerf, medical doctor specializing in endocrinology and metabolic diseases, Institut Pasteur de Lille
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2011-A00364-37
Record Dates: First submitted 2011-09-13; First posted 2011-11-29 (Estimated); Last update posted 2013-08-05 (Estimated); Status verified 2013-08

CONDITIONS: Age-related Macular Degeneration
Keywords: eggs; Optical Macular Pigment; Age Macular Degeneration; study for the Age Macular Degeneration prevention
MeSH Terms: conditions — Macular Degeneration | interventions — Nutritional Status

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- rich-eggs (Experimental): subjects consume 2 eggs rich in lutein/zeaxanthin and DHA per day during 4 months
  Interventions: Other: Nutritional study
- standard eggs (Active Comparator): subjects consume 2 standard eggs per day
  Interventions: Other: Nutritional study

INTERVENTIONS:
Other: Nutritional study — subjects consume 2 eggs per day during 4 months

SUMMARY:
This study is to determine the impact of the consumption of eggs rich in lutein/zeaxanthin from lucerne protein concentrate and DHA from microalgae on the plasma levels of these compounds but also on the macular pigment optical density, whose elevation may be beneficial in the prevention of Age-related Macular Degeneration (AMD).

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects (male or female),
* 18 to 55 years
* Having signed the consent form,
* Susceptible to accept the stresses generated by the study,
* Insured.

Exclusion Criteria:

* Corrected Visual Acuity <8/10th,
* History of cardiovascular disease, specifically coronary heart disease,
* Characterized dyslipidemia

  * Total cholesterol ³ 2.50 g / L, and / or triglycerides ³ 2.00 g / L
* Lipid-lowering treatment,
* Current smoking or person who stopped smoking less than 6 months
* Cataract or cataract surgery,
* Diabetes
* Body Mass Index (BMI)> 30 kg/m2,
* Taking food supplements in the 3 months preceding the start of the study (carotenoids, omega-3 fatty acids, phytosterols),
* Regular consumption in the three months preceding the start of the study products with added phytosterols.
* Regular consumption of high fatty fish or shellfish rich in omega-3 (4x a week or more): salmon, sardines, mackerel, herring, trout, tuna, red mullet, sea bass, bream, farmed turbot, mussels, squid / squid, anchovies.
* Allergy to eggs
* Dieting
* Difference significant weight over the last 3 months (> 3 kg)
* Inability to understand or adhere to the protocol
* Persons deprived of liberty
* People in a position to judicial protection
* Pregnant Women.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2011-10; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
change from baseline in optical density of macular pigment after 4 months of eggs consumption | before the eggs consumption and four months afterwards
  optical density of macular pigment was measured with a Heidelberg Retinal Angiograph (HRA)specially modify for the measure of the pigment.

SECONDARY OUTCOMES:
change from baseline in lutein and zeaxanthin in plasma and lipoproteins after 4 months of egg consumption | before the eggs consumption and four months afterwards
  lutein and zeaxanthin were measured by HPLC
change from baseline in fatty acids in plasma and lipoproteins after 4 months of egg consumption | before the eggs consumption and four months afterwards
  Fatty acids were measured by Gas Chromatography.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Michel Lecerf, MD, Principal Investigator — Institut Pasteur de Lille
Locations (1):
- Institut Pasteur de Lille, Lille, France